CLINICAL TRIAL: NCT00637429
Title: Human Immunodeficiency Virus (HIV) and Hepatitis B Virus (HBV) co-Infection and Liver Disease
Brief Title: HIV-HBV Co-Infection and Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Centre for Clinical Research Excellence in Infectious Diseases, Parkville (Unknown); Gilead Sciences (Industry)
Responsible Party: Professor Sharon Lewin, The Alfred Hospital and Monash University
Other Study IDs: ALF-263/06
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infections; HIV-HBV Co-Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General Co-infection: Individuals with HIV infection and hepatitis B surface antigen positive results who are currently receiving or planning to commence HAART.

SUMMARY:
Human immunodeficiency virus/Hepatitis B virus (HIV/HBV) co-infections are frequently observed due to shared routes of transmission, with reported figures indicating 6-9% of HIV-infected individuals in developed countries are chronically infected with HBV. HIV infection impacts on the natural progression of HBV infection, increasing levels of HBV replication and the risk of liver-associated mortality. Liver diseases associated with HBV are affected by the antiviral drugs used for HIV infection (toxic side effects), the current immune function in the patient, by improvements in the immune system brought about by control of the HIV infection, and by the development of resistance to the antiviral agents used for both the hepatitis B and the HIV infection. Co-infection with HBV increases the risk for hepatotoxicity in those individuals receiving highly active antiretroviral therapy (HAART) for their HIV infection.

This study will recruit patients who are co-infected with HIV and HBV, and are currently taking or who are about to commence HAART. The study cohort will include HIV-HBV co-infected individuals from the Alfred Hospital, the Royal Melbourne Hospital and high case load GP clinics who are referred to the Alfred Hospital.

The aim of the study is to investigate chronic hepatitis B and its impact on the progression of liver disease in HIV-infected persons receiving HAART.

This will be achieved by 6 monthly assessment with medical history, physical examination, bloods for markers of liver disease and hepatitis B activity and completion of questionnaires to measure adherence and alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* HIV positive
* 2 positive Hepatitis B surface antigen results 6 months apart
* provision of informed consent

Exclusion Criteria:

* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-HBV co-infected individuals from the Alfred Hospital, the Royal Melbourne Hospital and high case load GP clinics who are referred to the Alfred Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2007-11

PRIMARY OUTCOMES:
To investigate the efficacy and sustainability of HBV-active HAART on hepatitis B suppression by measuring changes in the HBV DNA levels as well as monitoring ALT levels, CD4 counts and HBV serology results. | 6 monthly assessment for 5 years

SECONDARY OUTCOMES:
The surveillance of antiviral resistance mutations that may develop in those individuals who are unable to sustain hepatitis B suppression | 6 monthly assessment for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Lewin, MD, PhD, Principal Investigator — The Alfred Hospital, Melbourne & Monash University
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia